Protocol Title, "Pain Outcomes After Anterior Cruciate Ligament Reconstruction with Posterior Capsular Marcaine Injection"

Cedars IRB # Pro41651

NCT # 02826551

Statistical Analysis Plan

Based on previous studies, the Mann-Whitney U test will check differences between numeric variables. Nonparametric Kruskal-Wallis tests can compare the analgesia level in the two groups and if possible ANOVA test can compare the analgesia duration. Chi-square tests will be utilized for any potential complications which will also be recorded. (J Inj Violence Res. 2013 Jun; 5(2): 84-88.) (Acta Ortop Bras. 2012;20(5); 285-90)

**Power Analysis** 

Prelim Power Analysis per STATS department @ Cedars: sample sizes of 26 for each group (N1=N2=26) = Total 52 patients to achieve 80% power to reject the null hypothesis of equal means when the population mean difference is 2 with a standard deviation for both groups of 2.5 and with a significance level (alpha) of 0.050 using a two-sided two-sample equal-variance t-test. A total of 60 patients will be enrolled to ensure we achieve adequate power for the study.